CLINICAL TRIAL: NCT02090816
Title: Combined Liver and Right Lung Resection for Colorectal Metastases by Means of J-shaped Thoracophrenolaparotomy
Status: Completed | Type: Observational
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Prof. Guido Torzilli, Professor of Surgery, University of Milan
Other Study IDs: Liver-lung-001
Record Dates: First submitted 2014-02-04; First posted 2014-03-18 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Colon Cancer Liver Metastasis; Multiple Pulmonary Nodules
MeSH Terms: conditions — Multiple Pulmonary Nodules

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Surgery of liver and lung: Patients carriers of both liver and right lung metastases in the same time
  Interventions: Procedure: Surgery of liver and lung

INTERVENTIONS:
Procedure: Surgery of liver and lung — Simultaneous resection of liver and right lung metastases in a single surgical session through a new approach

SUMMARY:
The purpose of this study is to determine whether J-shaped thoracophrenolaparotomy is effective in the surgical treatment of simultaneous liver and right lung metastases from colorectal cancer

DETAILED DESCRIPTION:
Right-sided lung metastases are resected synchronously with liver metastases by means of a thoracophrenolaparotomy.

The pre-operative staging includes for all patients colonoscopy, thoracic and abdominal contrast enhanced computed tomography (CT), contrast enhanced magnetic resonance (MRI) of the upper abdomen, and 18-fluorodeoxyglucose PET scan.

Laboratory examinations including liver function tests, spirometry, cardiologic and anesthesiological evaluation are also performed in alla patients.

Surgical Procedures The patient is placed in supine position with the arms extended laterally. The anaesthesiologist for selective lung insufflation positions the double lumen endotracheal tube. The J-shaped abdominal incision conventionally adopted for liver surgery is performed. In case of tumors involving segment 1 or cranial segment portion of segments 4 superior, 7 and 8 close to the caval confluence, the incision is prolonged along the 9th right intercostal space allowing the access to thoracic cavity. The incision of the skin and the external oblique muscle reaches the anterior axillary line. A small portion, about 2 centimetres, of the cartilaginous costal arch is removed, and then the diaphragm is divided in a radial direction. The inner parietal incision, involving parietal pleura and intercostal muscles is prolonged up to the posterior axillary line preserving the intercostal neurovascular bundle.

Intraoperative ultrasound (IOUS) is performed in all patients to stage the liver involvement as well as to assess the relation between tumors and vascular structures and guidance in the dissection of hepatic parenchyma. If nodules are isoechoic in comparison to the surrounding tissue, the staging is completed with contrast-enhanced IOUS (CEIOUS); the contrast agent consists of 4.8 mL of microbubbles filled with sulfur hexafluoride (SonoVue®; Bracco Imaging, Italy), which is injected intravenously.

Once surgical strategy is defined, the liver mobilization is completed by dividing the right and/or left triangular and coronary ligaments as needed. For combining the abdominal and thoracic procedures the right liver has to be mobilized at least up to the exposure of the inferior vena cava allowing larger radial incision of the diaphragm and enlarged view field to the thoracic cavity.

At first the thoracic surgeon performs the pulmonary part. The bed is tilted to the left side and exposure of right thoracic cavity is gained to the entire lung and the lateral mediastinum. With deflation and gentle retraction of the ipsilateral lung, the mediastinum and pericardium are exposed. Pulmonary ligament and lobar fissures are divided as needed. Manual palpation of the lung to detect the metastatic lesion is carried out. Then, wedge resection of the lung metastases is performed by using disposable stapler. Allowing the lung to collapse facilitates application of the stapling device and achievement of an adequate margin. Absorbable monofilament sutures are used, if necessary, to ensure haemostasis and/or small air leaks.

The hepatic resection is then started. Briefly, definition of the resection area with the main purpose of surrounding the tumor at its deepest portion combining the minimal parenchymal sacrifice and the flattest cut surface is performed under IOUS guidance. The hilar pedicle is then encircled with a tourniquet if dissection is not intended. Otherwise, in case of major hepatectomy, hilar dissection is performed. For all patients, parenchymal transection is obtained under intermittent clamping by Pringle maneuver continued for 15 minutes followed by 5 minutes of reperfusion without preconditioning. After 4 clamping cycles, reperfusion time is prolonged for 10 minutes. Liver dissection is accomplished using crush clamping technique, ligating with sutures all the vessels but those thinner which are coagulated using bipolar electrocautery . Before abdominal closure, the cut surface of the liver is sealed with haemostatic agent.

Closed suction abdominal drains are inserted in every patient around the liver, in variable number depending to the number and the size of liver cut surfaces. They are removed on the 7th postoperative day (POD) if the bilirubin level in the drain discharge sampled routinely on the 3rd, 5th, and 7th POD showed a decrement, and in any case was below 10 mg/ml.

One or two chest tube are placed in the pleural cavity, being removed from the 3rd POD, in absence of air leak within the bottle and if the serous output is below 200 mL/24h.

The ribs are approximated with pericostal sutures using braided absorbable sutures size 2. The diaphragm is closed with a single layer running suture. Peritoneum and fasciae of the chest and abdominal wall are closed in an anatomic pattern. Subcutaneous layer and skin are finally closed in the routine manner.

ELIGIBILITY:
Inclusion Criteria:

* Controlled primary disease;
* No extrahepatic lesion other than resectable pulmonary metastases at preoperative investigation;
* No lymph-node metastases except for those eventually present at the hepatic hilum;
* Disregarding number and distribution of liver metastases, technical resectability leaving at least a remnant liver volume of at least 40% of the total liver volume (calculated excluding the tumoral volume) featured by preserved inflow, outflow and biliary drainage. Zero mm free margin was considered acceptable in case of contact or close adjacency (< 5 mm) with 1st or 2nd order portal pedicles and/or major hepatic veins at their caval confluence;
* Disregarding number and distribution of lung metastases, all of the detected nodules could be completely removed preserving enough functioning remnant lung based on the results of the preoperative cardio-pulmonary functional tests;
* Patients eligible for a J-shaped thoracophrenolaparotomy because carrier of liver metastases located at the caval confluence, or in the paracaval portion of segment 1 or in the upper right segments (4 superior, 7 and 8), or presenting strong-adhesion or infiltration of the diaphragm.

Exclusion Criteria:

* Patients not suitable for surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tertiary care clinic
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2004-09; Primary Completion 2013-04 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Number of metastases removed | Baseline: date of surgical operation
  Evaluation of the resectability of whole metastases in liver and right lung in the same operation by means of the same surgical incision (J-shaped thoracophrenolaparotomy)

SECONDARY OUTCOMES:
Number of patients that received interventional treatments after surgery | Participants will be followed from the baseline (date of surgery) to 90 days after the operation
Number of re-operated patients | Participants will be followed from the baseline (date of surgery) to 90 days after the operation

CONTACTS AND LOCATIONS:
Overall Officials: Guido Torzilli, MD PhD FACS, Principal Investigator — University of Milan
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milan, Italy